CLINICAL TRIAL: NCT06764628
Title: An Open-label, Single-arm, Multicenter Phase I/II Clinical Study of SHR-4375 Injection in Patients With Advanced Solid Tumors to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy
Brief Title: A Study of SHR-4375 in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4375-101
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: SHR-4375

INTERVENTIONS:
Drug: SHR-4375 — SHR-4375 injection

SUMMARY:
This is an open-label, three-part study to evaluate the safety and efficacy of SHR-4375 for injection in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the ICF.
2. Measurable disease, as defined by RECIST v1.1.
3. The Eastern Cancer Cooperative Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 12 weeks.
5. Subjects with cytologically or histologically confirmed advanced solid tumors who have failed or are intolerant to standard therapy, have no standard therapy, or refuse standard therapy.

Exclusion Criteria:

1. Symptomatic, untreated or active central nervous system metastases.
2. With any active autoimmune disease or history of autoimmune disease.
3. Patients with active hepatitis B or hepatitis C.
4. Severe infections prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From Day 1 to 90 days after last dose.
Dose limiting toxicity (DLT) | From Day 1 to 12 months.
Maximal tolerable dose (MTD) | From Day 1 to 12 months.
Recommended phase 2 dose (RP2D) | From Day 1 to 12 months.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From Day 1 to 12 months.
Objective response rate (ORR) | From Day 1 to 12 months.
Disease control rate (DCR) | From Day 1 to 12 months.
Duration of response (DOR) | From Day 1 to 12 months.
Overall survival (OS) | From Day 1 to 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided